CLINICAL TRIAL: NCT05494099
Title: Extended Endoscopic Approaches to Non-malignant Maxillary Sinus Lesions Comparative Study
Brief Title: Extended Endoscopic Approaches to Non-malignant Maxillary Sinus Lesions Comparative
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eslam Mohamed Shata, doctor, Tanta University
Other Study IDs: maillary sinus approaches
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Maxillary Sinus Disease; Approach-Approach Conflict
Keywords: maxillary sinus; endoscopic approaches

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A (1st 25 patients): The middle meatal mega-antrostomy approach.
  Interventions: Procedure: endoscopic maxillary mega-antrostomy
- Group B (2nd 25 patients): The endoscopic modified medial maxillectomy approach.
  Interventions: Procedure: Endoscopic Modified Medial Maxillectomy
- Group C (3rd 25 patients): The endoscopic prelacrimal recess approach.
  Interventions: Procedure: Modified endoscopic pre-lacrimal approach

INTERVENTIONS:
Procedure: endoscopic maxillary mega-antrostomy — a mucosal sparing technique that facilitates mucus clearance and sinus irrigation in terminally dysfunctional maxillary sinuses. EMMA involves extending the antrostomy through the posterior half of the inferior turbinate down to the floor of the nose, creating a significantly enlarged antrostomy.
  Groups: Group A (1st 25 patients)
Procedure: Endoscopic Modified Medial Maxillectomy — In this approach, the maxillary sinus is operated upon, while the inferior turbinate and nasolacrimal duct are preserved.
  Groups: Group B (2nd 25 patients)
Procedure: Modified endoscopic pre-lacrimal approach — The approach involves making a curved mucosal incision on the lateral nasal wall just anterior to the head of the inferior turbinate. The nasal mucosa was then undermined off the lateral nasal wall. The maxillary sinus was entered with a chisel, and the medial bony wall of the maxillary sinus removed.
  Groups: Group C (3rd 25 patients)

SUMMARY:
The aim of this study is to compare the outcomes of endoscopic middle meatus mega-antrostomy, endoscopic pre-lacrimal recess approach and endoscopic modified medial maxillectomy regarding: 1.Assessment of the accessibility of each approach to visualize and reach the different walls and recesses of the maxillary sinus. 2. Any intraoperative or postoperative complications. 3. Any post-operative recurrence or residue detected by endoscopic examination. 4. Symptomatic relief by pre- and post-operative Sino-Nasal Outcome Test 22, Arabic translation and validation (SNOT-22) which is a reliable and valid outcome measure for CRS patients.

DETAILED DESCRIPTION:
A wide range of surgical ways to reach maxillary sinus. Historically, maxillary sinus was entered by external approaches such as lateral rhinotomy etc. in benign or malignant diseases, but now endoscopic approaches have recently replaced external approaches as the standard of treatment of maxillary sinus diseases due to reduced morbidity, improved visualisation and low recurrence rates of benign tumours.

Studies found that middle meatal antrostomy only provided access to about 24-34 percent of the total sinus volume only and rarely offer access to the anterior wall and sinus floor, regardless of the angled instruments used .Endoscopic maxillary mega-antrostomy is typically used as a revision procedure in patients with maxillary sinusitis refractory to surgery. The resulting antrostomy is greatly enlarged and allows the sinus to drain more easily by gravity, as well as admitting topical therapy more readily .

Radical endoscopic medial maxillectomy is indicated for the resection of benign and malignant sinonasal neoplasms when wide surgical access and tumor clearance is required However, resection of the inferior turbinate head may contributes to nasal crusting, dryness and empty nose syndrome ,so modified endoscopic medial maxillectomy gives better access to the maxillary sinus, with preserving the head of the inferior turbinate Pre-lacrimal recess approach allows for direct access to the sinus with 0-degree endoscopes and straight instruments, and thus improved visualisation of its contents especially anterior sinus wall, better handling of tools with preservation of inferior turbinate and nasolacrimal duct It is difficult to select suitable approach to maxillary sinus to ensure proper intraoperative visualization and better access to disease with fewer complications that is why we do this study.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory disease of the maxillary sinus in the context of allergic or infective rhinosinusitis, with or without formation of inflammatory polyps. When such cases fail to respond to maximal medical therapy.
* Benign and locally malignant neoplasms of the maxillary sinus (ex: inverted papilloma) which are planned to be removed by extended endoscopic approach.

Exclusion Criteria:

* Patients who are unfit to surgery (ex: with bleeding disorders or severe systemic diseases).
* Patients who refuse surgery or difficult to be followed up.
* Patients with minimal lesions who respond to medical treatment.
* Patients with malignant tumor of maxillary sinus proved by histopathology.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic rhinosinusitis who not respond to medical treatment and are planned to be operated by endoscopic sinus surgery.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Intra-operative Endoscopic Assesment | Intraoperative only
  Assessment of the accessibility of endoscopic approach which will be evaluated by using different types of telescopes to visualize and reach the different walls and recesses of the maxillary sinus

SECONDARY OUTCOMES:
Sino-Nasal Outcome Test 22,. Arabic translation and validation (SNOT-22) | 3 months
  Assess the effect of each endoscopic approach on recurrence rate of maxillary sinus lesions.
  regular endoscopic examination first visit after one week, second after 3 weeks and the third after 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Mu Hegazy, MD, Study Director — Tanta University Hospital, Egypt.; Ahmed Mo Gamea, MD, Study Director — Tanta University Hospital, Egypt.; Mohamed Os Tomom, MD, Study Director — Tanta University Hospital, Egypt.
Locations (1):
- Faculty of medicine, Tanta, Gharbia Government, Egypt

IPD SHARING:
Plan to Share IPD: Yes
To compare the outcomes of endoscopic middle meatus mega-antrostomy, endoscopic pre-lacrimal recess approach and endoscopic modified medial maxillectomy regarding: 1.Assessment of the accessibility of each approach to visualize and reach the different walls and recesses of the maxillary sinus. 2. Any intraoperative or postoperative complications. 3. Any post-operative recurrence or residue detected by endoscopic examination. 4. Symptomatic relief by pre- and post-operative SNOT-22 which is a reliable and valid outcome measure for CRS patients.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year

REFERENCES:
- [Background] Goudakos JK, Blioskas S, Nikolaou A, Vlachtsis K, Karkos P, Markou KD. Endoscopic Resection of Sinonasal Inverted Papilloma: Systematic Review and Meta-Analysis. Am J Rhinol Allergy. 2018 May;32(3):167-174. doi: 10.1177/1945892418765004. Epub 2018 Apr 12. PMID 29649889
- [Background] Robey A, O'Brien EK, Leopold DA. Assessing current technical limitations in the small-hole endoscopic approach to the maxillary sinus. Am J Rhinol Allergy. 2010 Sep-Oct;24(5):396-401. doi: 10.2500/ajra.2010.24.3486. PMID 21244743
- [Background] Cho DY, Hwang PH. Results of endoscopic maxillary mega-antrostomy in recalcitrant maxillary sinusitis. Am J Rhinol. 2008 Nov-Dec;22(6):658-62. doi: 10.2500/ajr.2008.22.3248. PMID 19178809
- [Background] Woodworth BA, Parker RO, Schlosser RJ. Modified endoscopic medial maxillectomy for chronic maxillary sinusitis. Am J Rhinol. 2006 May-Jun;20(3):317-9. doi: 10.2500/ajr.2006.20.2850. PMID 16871936
- [Background] Gosau M, Rink D, Driemel O, Draenert FG. Maxillary sinus anatomy: a cadaveric study with clinical implications. Anat Rec (Hoboken). 2009 Mar;292(3):352-4. doi: 10.1002/ar.20859. PMID 19248167
- [Background] Sadeghi N, Al-Dhahri S, Manoukian JJ. Transnasal endoscopic medial maxillectomy for inverting papilloma. Laryngoscope. 2003 Apr;113(4):749-53. doi: 10.1097/00005537-200304000-00031. PMID 12671441
- [Background] Wormald PJ, Ooi E, van Hasselt CA, Nair S. Endoscopic removal of sinonasal inverted papilloma including endoscopic medial maxillectomy. Laryngoscope. 2003 May;113(5):867-73. doi: 10.1097/00005537-200305000-00017. PMID 12792324
- [Background] Luong A, Citardi MJ, Batra PS. Management of sinonasal malignant neoplasms: defining the role of endoscopy. Am J Rhinol Allergy. 2010 Mar-Apr;24(2):150-5. doi: 10.2500/ajra.2010.24.3451. PMID 20338116
- [Background] Kastl KG, Rettinger G, Keck T. The impact of nasal surgery on air-conditioning of the nasal airways. Rhinology. 2009 Sep;47(3):237-41. doi: 10.4193/Rhin08.014. PMID 19839243
- [Background] Dayal A, Rhee JS, Garcia GJ. Impact of Middle versus Inferior Total Turbinectomy on Nasal Aerodynamics. Otolaryngol Head Neck Surg. 2016 Sep;155(3):518-25. doi: 10.1177/0194599816644915. Epub 2016 May 10. PMID 27165673
- [Background] Morrissey DK, Wormald PJ, Psaltis AJ. Prelacrimal approach to the maxillary sinus. Int Forum Allergy Rhinol. 2016 Feb;6(2):214-8. doi: 10.1002/alr.21640. Epub 2015 Sep 8. No abstract available. PMID 26346189